CLINICAL TRIAL: NCT04905511
Title: Preliminary Safety of The TRUE Vascular Graft for Hemodialysis Access (TRUE HD I Study)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vascudyne, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP-001
Record Dates: First submitted 2021-05-21; First posted 2021-05-27 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: Prospective, nonrandomized, single-arm, single-center, open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- TRUE Vascular Graft (Experimental): Patients will be implanted with the TRUE Vascular Graft in the upper arm or forearm
  Interventions: Biological: natural human collagen arteriovenous graft for hemodialysis access

INTERVENTIONS:
Biological: natural human collagen arteriovenous graft for hemodialysis access — The True Vascular Graft will be implanted in the forearm or upper arm in a straight or curved configuration.

SUMMARY:
Prospective, nonrandomized, single-arm, single-center, open-label, first-in-human clinical study in subjects with end-stage renal disease (ESRD) and not candidates for an autogenous fistula creation.

DETAILED DESCRIPTION:
Prospective, nonrandomized, single-arm, single-center, open-label, first-in-human clinical study in subjects with end-stage renal disease (ESRD) and not candidates for an autogenous fistula creation. Subjects will be followed regularly with office visits at the investigational site at days 15, 29, 57 and weeks 12, 26 for vessel imaging, blood draws and other follow-up tests.

ELIGIBILITY:
Inclusion Criteria:

* Patients with end stage renal disease (ESRD) who are not, or who are no longer, candidates for creation of a simple autogenous AV fistula (radio-cephalic or brachio-cephalic without requiring transposition) and therefore need placement of an AV graft in the upper extremity to start or maintain hemodialysis therapy.
* Either on hemodialysis or expected to start hemodialysis within 12 weeks of study conduit implantation.
* Patients between 18 and 75 years old, inclusive.
* Life expectancy of at least 1 year.
* Negative COVID-19 test within 3 days prior to surgery and negative for symptoms within 14 days prior to surgery.
* Able to communicate meaningfully with investigative staff and able to comply with entire study procedures.
* Willing and competent to give written informed consent.

Exclusion Criteria:

* History or evidence of severe cardiac disease (NYHA Functional Class III or IV), myocardial infarction within six months prior to study entry (Day 1), ventricular tachyarrhythmias requiring continuing treatment, or unstable angina.
* Uncontrolled or poorly controlled diabetes; hospitalization for poor glucose control within the previous 6 months.
* History or evidence of severe peripheral vascular disease in the upper limbs
* Known or suspected central vein obstruction on the side of planned graft implantation.
* Documented hypercoagulable state or history of thromboembolic events or history of repeated venous catheter clotting.
* Known Positive COVID 19 test result or known exposure to COVID 19 in past 4 months.
* Known active infection including dental infection, osteomyelitis and other conditions which could present a local or systemic risk of infection.
* Bleeding diathesis.
* Contraindication to or known serious allergy to anticoagulant, aspirin, or planned antiplatelet therapy. History of heparin-induced thrombocytopenia.
* Contraindication to or known serious allergy to penicillin.
* Ongoing therapy with vitamin K antagonists or direct thrombin inhibitors or factor Xa inhibitors.
* Immunodeficiency including AIDS / HIV or active autoimmune disease, or on immunosuppressant therapy.
* Previous PTFE graft in the operative limb unless the TRUE graft can be placed more proximally than the previous failed graft.
* More than 1 failed PTFE graft in the operative limb.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 10 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Safety, adverse events | 26 weeks
  incidence of clinically significant aneurysm, anastomotic bleeding, graft or anastomotic rupture, graft infection, and implant site irritation, inflammation, or infection
Patency | 26 weeks
  time to loss of patency from implantation by Kaplan Meier

SECONDARY OUTCOMES:
Immunology | baseline through 4 weeks
  assess changes in panel reactive antibody (PRA) from baseline
Intervention rate | through 26 weeks
  rate of interventions needed to maintain patency

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Ebner, MD, Principal Investigator — Sanatorio Italiano
Locations (1):
- Sanatario Italiano, Asunción, Paraguay

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Syedain ZH, Graham ML, Dunn TB, O'Brien T, Johnson SL, Schumacher RJ, Tranquillo RT. A completely biological "off-the-shelf" arteriovenous graft that recellularizes in baboons. Sci Transl Med. 2017 Nov 1;9(414):eaan4209. doi: 10.1126/scitranslmed.aan4209. PMID 29093182